CLINICAL TRIAL: NCT03513159
Title: Transsectoral Intervention Program for Improvement of Geriatric Care in Regensburg
Brief Title: Improvement of Transition From Hospital to Home for Older Patients in Germany
Acronym: TIGER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Hospital of the Order of St.John of God Regensburg, Barmherzige Brueder, Germany (Unknown); Regensburg Physicians Network RAEN (Unknown); Friedrich-Alexander-Universität Erlangen-Nürnberg (Other); AOK Bayern (Industry); Institute for Nursing Sciences, University of Bielefeld, Germany (Unknown); Federal Association for Geriatrics, Germany (Unknown); Federal Joint Committee (Other Government); Institute for Community Medicine, University of Greifswald, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IBA-2018-TIGER
Record Dates: First submitted 2018-04-17; First posted 2018-05-01 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Geriatric Patients in the Transition From Hospital to Home
Keywords: transitional care, geriatric, readmission,; discharge; quality of life

STUDY DESIGN:
Intervention Model Description: The Intervention Group will be supported by the activities of the pathfinder, the Control Group will not. Both Groups will be tested for functional and nutritional Status and for Quality of life and stress scores.
Masking Description: The patients data will be anonymized and entered into an electronic Case Report form. The Outcomes Assessor will only see the anonymized data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pathfinder support (Experimental): Pathfinder support with development of an individual care plan for the intervention patients and their informal caregivers, with the hospital physicians already inside the hospital setting. This will then be developed and improved further during up to twelve months after hospital release with the primary physician. The pathfinders will coordinate the ambulatory care team services and closely involve the primary physicians. The patients and their informal caregivers will be empowered and educated to achieve a stabilization or improvement in functionality, independence, quality of life, coping with disease, nutritional status and wound healing process. In the regular assessments they will be tested for functionality and nutritional parameters, quality of life and stress scores.
  Interventions: Behavioral: Pathfinder support
- Control without pathfinder support (No Intervention): Control patients will not be supported by pathfinders. In regular assessments they will be tested for functionality and nutritional parameters, quality of life and stress scores.

INTERVENTIONS:
Behavioral: Pathfinder support — A pathfinder will support the patient with structured activities.
  Arms: Pathfinder support

SUMMARY:
The aim of the transsectoral care project TIGER is the reduction of readmission rates of geriatric patients. This aim shall be achieved by improving the hitherto inadequate care process for geriatric patients in the transition from hospital to home. The program offers substantial support of patients and their informal caregivers in the transition process from hospital to home via so called pathfinders, specialized nurses in geriatrics.The pathfinders effectively intertwine stationary and ambulatory care teams caring for a patient, thereby augmenting and complementing effective hospital release management.

DETAILED DESCRIPTION:
Especially for older, chronically ill persons, a hospital stay can promote significant losses in functionality, independence and quality of life, and can increase nutrition deficits and the risk for infections, leading to the occurrence of severe gaps in care after hospital release and to an increased risk for readmission rates.

Even if the German government has recognized the necessity of a multiprofessional integrated care program for older, vulnerable patients and has installed a hospital release management program situated in hospitals in 2012, clarifying entitlements to benefits and setting up ambulatory services contacts, this does not yet meet the complex needs of geriatric patients and their informal caregivers.

Internationally, the Transitional Care Model (TCM) has been developed (M. Naylor et al. 1994) to address the deficits in care of older patients in transition between hospital to home. Via a series of defined activities, a disruption of the care supply chain for older patients in this transition process is being avoided.

The TIGER program will address the needs of geriatric patients and their informal caregivers and will support them via structured continuous activities, on the basis of the TCM, by so called pathfinders, nurses specialized in geriatrics. These pathfinders will develop an individual care plan with the patients, their informal caregivers and the hospital physicians already inside the hospital setting and will then develop and improve this further during up to twelve months after the hospital release of the patient. The pathfinders will coordinate the ambulatory care team services and closely involve the primary physicians. The patients and their informal caregivers will be empowered and educated to achieve a stabilization or improvement in functionality, independence, quality of life, coping with disease, nutritional status and wound healing process of the patients.

The aim of the program is that these activities will lead to a reduction of necessary readmission rates of geriatric patients.

Efficacy, practicability, and limitations of the program will be evaluated scientifically and economically and will be analyzed for a possible saving of costs for the health care system.

ELIGIBILITY:
Inclusion Criteria:

will go back home after Hospital stay, AOK Patient, MiniMentalStateExamination MMSE score of at least 22, is living within 50 km range of the hospital

Exclusion Criteria:

palliative status, planned readmission into hospital within next 4 weeks

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 252 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Readmission Rate | up to 12 months
  The number of readmissions of a patient into a hospital within up to 15 months (study period for the patient.plus 3 months prior to enrollment).

SECONDARY OUTCOMES:
Functionality and mobility - 1 | up to 12 months
  Timed up and Go in seconds
Functionality and mobility - 2 | up to 12 months
  Instrumental activities of daily living (IADL) in scale
Functionality and mobility - 3 | up to 12 months
  handgrip strength in kilogramms
Functionality and mobility - 4 | up to 12 months
  pedometer activPAL3 micro
Functionality and mobility - 5 | up to 12 months
  Short physical performance battery (SPPB) in scale
Nutritional status | up to 12 months
  measured bei Mini Nutritional Assessment (MNA)
Health-related quality of life | up to 12 months
  Measured by Short-Form-Health Survey (SF-12) questionnaire in scale
Depression | up to 12 months
  Measured by Geriatric Depression Scale (GDS) in scale
Cognitive Status - 1 | up to 12 months
  Measured by Mini-Mental State Examination (MMSE) in scale
Cognitive Status - 2 | up to 12 months
  Trail Making Test A&B in seconds
Burden of informal caregivers - 1 | up to 12 months
  Measured by Zarith-questionnaires in scale
Burden of informal caregivers - 2 | up to 12 months
  Perceived Stress Questionnaire (PSQ)-questionnaires in scale
Transfers into nursing homes | Up to 12 months
  Comparison between intervention and control group. Data made available by cooperating partner Allgemeine Ortskrankenkasse (AOK) sickness fund in percent
Care situation, care supply and quality of care at home | up to 12 months
  Measured by Neues BegutAchtungsinstrument (NBA, Buscher, Wingenfeld & Schaeffer, 2011) as scale

CONTACTS AND LOCATIONS:
Overall Officials: Cornel Sieber, Prof. Dr., Study Director — Institute for Biomedicine of Aging
Locations (2):
- Germany (2):
  - Hospital of the Order of St.John of God Regensburg, Regensburg, Bavaria
  - Institute for Biomedicine of Aging, University of Erlangen-Nürnberg, Nuremberg

IPD SHARING:
Plan to Share IPD: Yes
The final anonymized trial data set will be available to the TIGER consortium. After completion of evaluation and dissemination by the TIGER-consortium, the goal is that an anonymized data set will be made available to interested Researchers upon reasonable request, being deposited in a repository of the University.
  During finalization of the study a detailed data sharing plan will be developed and introduced into this trial registry.
Supporting Information: Study Protocol, CSR
Time Frame: The repository of the data set is under construction with the University.
Access Criteria: Anonymized data set will be available to interested Researchers upon reasonable request

REFERENCES:
- [Derived] Gehr TJ, Freiberger E, Sieber CC, Engel SA. A typology of caregiving spouses of geriatric patients without dementia: caring, worried, desperate. BMC Geriatr. 2021 Sep 6;21(1):483. doi: 10.1186/s12877-021-02425-1. PMID 34488636
- [Derived] Rimmele M, Wirth J, Britting S, Gehr T, Hermann M, van den Heuvel D, Kestler A, Koch T, Schoeffski O, Volkert D, Wingenfeld K, Wurm S, Freiberger E, Sieber C; TIGER consortium. Improvement of transitional care from hospital to home for older patients, the TIGER study: protocol of a randomised controlled trial. BMJ Open. 2021 Feb 8;11(2):e037999. doi: 10.1136/bmjopen-2020-037999. PMID 33558344